CLINICAL TRIAL: NCT03596775
Title: Effect of Single-dose Dexmedetomidine on Emergence Agitation and Postoperative Behavior Changes After Sevoflurane Anesthesia in Children
Brief Title: Effect of Dexmedetomidine on Emergence Agitation and Postoperative Behavior Changes in Children
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Jin Dong Liu, Principal Investigator, Xuzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XYFY-2018-0061
Record Dates: First submitted 2018-06-20; First posted 2018-07-24 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Emergence Agitation
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine group (Experimental): the children received 0.5 μg/kg of intravenous dexmedetomidine over 10 minutes after induction of anesthesia
  Interventions: Drug: Dexmedetomidine
- Control Comparator group (Placebo Comparator): the children received 10ml saline over 10 minutes after induction of anesthesia
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Dexmedetomidine — Children in Dexmedetomidine group receive intravenous dexmedetomidine 0.5 ug/kg over 10 minutes after induction of anesthesia.
  Arms: Dexmedetomidine group
Drug: saline — Children in Control Comparator group receive intravenous saline 10ml over 10 minutes after induction of anesthesia.
  Arms: Control Comparator group

SUMMARY:
Emergence agitation (EA) is a dissociated state of consciousness in which the child is inconsolable, irritable, uncooperative, typically thrashing, crying, moaning, or incoherent. Although usually transient, it is not only an extremely distressing event for children, parents, and staff, but may also result in self-injury or the need for restraint. The prevalence in children appears to be between 10% and 80% depending upon the definition and measurement tools used and is more frequently observed in the pre-school age-group. A clear correlation has been found between EA and negative postoperative behavioral changes, including anxiety, eating and sleeping disorders, enuresis, fear of darkness, that may persist for an extended period of time affecting emotional and cognitive development.Currently, numerous interventions have been studied to manage EA after surgery. Among them, dexmedetomidine (DEX) as a kind of highly selective α2 adrenergic receptor agonist has been done to reduce EA in children. Unfortunately, no studies examined posthospitalization negative behaviour changes.

DETAILED DESCRIPTION:
The high incidence of EA and postoperative behavioural changes has encouraged paediatric anaesthetists and researchers to study methods to improve the perioperative care of children. Dexmedetomidine is a selective alpha-2 receptor agonist with properties that make it attractive to pediatric use. It provides sedation and anxiolysis acting on these receptors in the locus ceruleus of the pons. It also exerts dose-dependent moderate primary analgesic effects through activation of alpha-2 adrenoreceptors in the dorsal spinal horn causing a subsequent decrease in substance P release. The study aims to explore whether a single low-dose dexmedetomidine in the perioperative period has a preventive effect on EA in children, and through short-term and long-term follow-up, to investigate the effect on post-hospitalization behavioural changes.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 2-7 years old
2. American Society of Anesthesiologists（ASA） score of I or II
3. Selective ear, nose, and throat surgery under general anaesthesia with sevoflurane

Exclusion Criteria:

1. Emergency surgery
2. were intubated before induction of anaesthesia or not planned for extubation after anaesthesia
3. had critical illness with haemodynamic instability, active bleeding, cancer, cardiac diseases including arrhythmias, malignant hyperthermia
4. intellectual disability, or neurological illness with agitation-like symptoms
5. weighed more than 50 kg
6. were allergic to dexmedetomidine
7. The use of sedative or analgesic medications before surgery

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of EA as assessed by the Pediatric Anesthesia Emergence Delirium (PAED) scale | within 30 minutes after extubation in the post-anaesthesia care unit
  Use the Pediatric Anesthesia Emergence Delirium (PAED) scale to record the incidence of EA.The score ranges from 0 to 20 points. A score of 10 or above is considered as EA.

SECONDARY OUTCOMES:
Pain scores as assessed by the Face, Legs, Activity, Cry, Consolability (FLACC) scale | within 30 minutes after extubation in the post-anaesthesia care unit
  Use the Face, Legs, Activity, Cry, Consolability (FLACC) scale to record the pain scores. The score ranges from 0 to 10 points. A score of 4 or above is considered as pain.
Rescue analgesia and sedative drug consumption | within 30 minutes after extubation in the post-anaesthesia care unit
  Rescue analgesia and sedative drug consumption in the post-anaesthesia care unit
Incidence of adverse events | within 30 minutes after extubation in the post-anaesthesia care unit
  Incidence of adverse events in the post-anaesthesia care unit
Post-hospitalization negative behaviour changes as assessed by the Post Hospitalisation Behaviour Questionnaire (PHBQ) scale | 1 day, 2 days,30 days post surgery
  Use the Post Hospitalisation Behaviour Questionnaire (PHBQ) scale to record the incidence of Post-hospitalization negative behaviour changes.This consists of 27 items describing six subscales: general anxiety, separation anxiety, sleep anxiety, eating disturbances, aggression against authority and apathy/withdrawal.The possible answers were provided on a scale from 1 to 5 ('much less', 'less', 'unchanged', 'more' or 'much more' than before hospitalisation).A score of 0 was awarded if no negative behaviour was reported either before or after surgery.Total score was calculated by adding up all responses.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Dong Liu, M.S, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data(IPD) will be available when this trial is finished and the article have been published

REFERENCES:
- [Background] Costi D, Cyna AM, Ahmed S, Stephens K, Strickland P, Ellwood J, Larsson JN, Chooi C, Burgoyne LL, Middleton P. Effects of sevoflurane versus other general anaesthesia on emergence agitation in children. Cochrane Database Syst Rev. 2014 Sep 12;2014(9):CD007084. doi: 10.1002/14651858.CD007084.pub2. PMID 25212274
- [Background] Pickard A, Davies P, Birnie K, Beringer R. Systematic review and meta-analysis of the effect of intraoperative alpha(2)-adrenergic agonists on postoperative behaviour in children. Br J Anaesth. 2014 Jun;112(6):982-90. doi: 10.1093/bja/aeu093. Epub 2014 Apr 11. PMID 24727829
- [Background] Tsiotou AG, Malisiova A, Kouptsova E, Mavri M, Anagnostopoulou M, Kalliardou E. Dexmedetomidine for the reduction of emergence delirium in children undergoing tonsillectomy with propofol anesthesia: A double-blind, randomized study. Paediatr Anaesth. 2018 Jul;28(7):632-638. doi: 10.1111/pan.13397. Epub 2018 May 12. PMID 29752853
- [Background] Silva LM, Braz LG, Modolo NS. Emergence agitation in pediatric anesthesia: current features. J Pediatr (Rio J). 2008 Mar-Apr;84(2):107-13. doi: 10.2223/JPED.1763. PMID 18372935
- [Background] Sun L, Guo R, Sun L. Dexmedetomidine for preventing sevoflurane-related emergence agitation in children: a meta-analysis of randomized controlled trials. Acta Anaesthesiol Scand. 2014 Jul;58(6):642-50. doi: 10.1111/aas.12292. Epub 2014 Mar 3. PMID 24588393
- [Background] Kain ZN, Caldwell-Andrews AA, Maranets I, McClain B, Gaal D, Mayes LC, Feng R, Zhang H. Preoperative anxiety and emergence delirium and postoperative maladaptive behaviors. Anesth Analg. 2004 Dec;99(6):1648-1654. doi: 10.1213/01.ANE.0000136471.36680.97. PMID 15562048